CLINICAL TRIAL: NCT02930330
Title: Interval Training in Cardiac Rehabilitation: Effects on Cardiorespiratory Fitness and Platelet Function - A Randomized Controlled Trial
Brief Title: Interval Training in Cardiac Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: Medical Scientific Fund of the Mayor of Vienna (Other); Austrian Heart Funds (Unknown)
Responsible Party: Principal Investigator, Stefan Heber, Dr. Med. Univ., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Heber 15136
Record Dates: First submitted 2016-10-07; First posted 2016-10-12 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Atherosclerosis; Coronary Artery Disease
Keywords: Exercise; Interval training; Blood platelets; Platelet function tests; Physical fitness; Rehabilitation
MeSH Terms: conditions — Atherosclerosis; Coronary Artery Disease; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interval (Experimental): 2x / week INT
  2x / week CONT
  Interventions: Behavioral: INT; Behavioral: CONT
- Continuous (Active Comparator): 4x / week CONT
  Interventions: Behavioral: CONT

INTERVENTIONS:
Behavioral: INT — * 5 min warm-up (40% Pmax*)
  * 30 min high intensity interval training (1 min 100% Pmax, 1 min 20% Pmax, in alternating sequence)
  * 10 min cool-down (30% Pmax)
  Pmax*: Maximal power output (Watt) achieved at the end of an incremental exercise test.
  Other Names: High intensity interval training
  Arms: Interval
Behavioral: CONT — * 5 min warm-up (40% Pmax*)
  * 30 min moderate intensity continuous training (60% Pmax)
  * 10 min cool-down (30% Pmax)
  Pmax*: Maximal power output (Watt) achieved at the end of an incremental exercise test.
  Other Names: Moderate intensity continuous training

SUMMARY:
The purpose of this study is to determine whether high intensity interval training (INT) is more effective in suppressing platelet reactivity than continuous, moderate intensity training (CONT) in patients undergoing cardiac rehabilitation after percutaneous coronary intervention.

DETAILED DESCRIPTION:
Background: Platelets play an important role in cardiovascular disease: First, they promote the development of atherosclerotic lesions, and second, platelets form vessel occluding thrombi on top of (ruptured) lesions, ultimately leading to thrombotic events like myocardial infarctions (MCI). Whereas acute, strenuous exercise causes platelet activation and transiently increases the risk for MCIs, long-term chronic exercise training results in a clear reduction of both platelet activation and MCI incidence.

Exercise training plays a key role in cardiac rehabilitation, since improvements in cardiorespiratory fitness (CRF) are associated with decreased mortality in these patients. With respect to CRF improvements, high-intensity interval training has been demonstrated to be more effective than moderate-intensity continuous exercise. However, the beneficial effect of high-intensity interval training on platelet function in patients with cardiovascular disease has never been investigated.

Scientific question: The aim of this study is to determine the effect of interval training in cardiac rehabilitation on platelet function.

Hypotheses: Cardiac rehabilitation with interval training components (INT) reduces

1. platelet activation and platelet reactivity at physical rest
2. changes of platelet activation and -reactivity induced by acute, strenuous exercise to a greater extent than cardiac rehabilitation consisting exclusively of moderate-intensity continuous exercise training (CONT).

Work program: 80 patients at the beginning of phase II cardiac rehabilitation will be randomly assigned to an interval group or to a control group. In both groups, patients will exercise 4x / week for 12 weeks. At the beginning, after 6 weeks and at the end an exercise test will be carried out. Blood will be taken before (platelet function at rest) and immediately after each exercise test (platelet function after acute, strenuous exercise). Basal platelet activation as well as platelet responsiveness towards a platelet agonist (platelet reactivity) will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* No regular exercise training within the last 6 months
* Dual anti-platelet therapy (low-dose aspirin plus ADP(adenosine diphosphate)-receptor antagonist)
* Status post percutaneous coronary intervention after recent acute coronary syndrome as underlying reason for current rehabilitation
* Eligibility for outpatient cardiac rehabilitation according to Table I in Niebauer et al. 2013 (PMID: 22508693)

Exclusion Criteria:

* Type II diabetes mellitus
* Aortic aneurysm / dissection
* Uncontrolled hypertension (>180/110 mmHg)
* Pulmonary hypertension (>55 mmHg)
* Previously known hereditary platelet disorders
* Disorders of plasmatic coagulation
* Anemia (Hb < 13g/dl)
* History of end-stage liver or kidney disease

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2015-10; Primary Completion 2017-06-14 (Actual); Study Completion 2017-06-14 (Actual)

PRIMARY OUTCOMES:
Platelet reactivity at physical rest: EC50 of TRAP-6 in terms of platelet CD62P expression. Unit of Measure: µM (Micromolar) | 6 weeks
  Platelet reactivity as measured by half maximal effective concentration (EC50) of the platelet agonist TRAP-6 (Thrombin receptor activating peptide-6; SFLLRN) in terms of platelet CD62P (P-selectin) expression, as described in Heber et al. 2016 (PMID: 26909532). The percentage of CD62P expressing platelets is quantified by flow cytometry without and with increasing concentrations of the platelet agonist TRAP-6. EC50 of TRAP-6 is estimated by fitting a four parameter logistic dose-response curve to flow cytometry data as a function of agonist concentration, aggregating multiple measurements to one reported value (EC50) with the unit µM.
  Treatment effects on platelet reactivity at physical rest after 6 weeks (INT vs. CONT) are estimated by ANCOVA, with baseline values as covariate.

SECONDARY OUTCOMES:
Platelet reactivity at physical rest: EC50 of TRAP-6 in terms of platelet CD62P expression. Unit of Measure: µM | 12 weeks
  Platelet reactivity as measured by half maximal effective concentration (EC50) of the platelet agonist TRAP-6 (Thrombin receptor activating peptide-6; SFLLRN) in terms of platelet CD62P (P-selectin) expression. The percentage of CD62P expressing platelets is quantified by flow cytometry without and with increasing concentrations of the platelet agonist TRAP-6. EC50 of TRAP-6 is estimated by fitting a four parameter logistic dose-response curve to flow cytometry data as a function of agonist concentration, aggregating multiple measurements to one reported value (EC50) with the unit µM.
  Treatment effects on platelet reactivity at physical rest after 12 weeks (INT vs. CONT) are estimated by ANCOVA, with baseline values as covariate.
Cardiorespiratory fitness: Maximal power output | 6 weeks
  Maximal power output (Watt / kg bodyweight) at the end of an incremental exercise test
Cardiorespiratory fitness: Maximal power output | 12 weeks
  Maximal power output (Watt / kg bodyweight) at the end of an incremental exercise test
Cardiorespiratory fitness: Maximal oxygen consumption | 6 weeks
  Maximal oxygen consumption (ml/min/kg bodyweight) at the end of an incremental exercise test
Cardiorespiratory fitness: Maximal oxygen consumption | 12 weeks
  Maximal oxygen consumption (ml/min/kg bodyweight) at the end of an incremental exercise test

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Heber, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- MUVienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Niebauer J, Mayr K, Tschentscher M, Pokan R, Benzer W. Outpatient cardiac rehabilitation: the Austrian model. Eur J Prev Cardiol. 2013 Jun;20(3):468-79. doi: 10.1177/2047487312446137. Epub 2012 Apr 16. PMID 22508693
- [Background] Heber S, Assinger A, Pokan R, Volf I. Correlation between Cardiorespiratory Fitness and Platelet Function in Healthy Women. Med Sci Sports Exerc. 2016 Jun;48(6):1101-10. doi: 10.1249/MSS.0000000000000882. PMID 26909532
- [Derived] Heber S, Fischer B, Sallaberger-Lehner M, Hausharter M, Ocenasek H, Gleiss A, Fischer MJM, Pokan R, Assinger A, Volf I. Effects of high-intensity interval training on platelet function in cardiac rehabilitation: a randomised controlled trial. Heart. 2020 Jan;106(1):69-79. doi: 10.1136/heartjnl-2019-315130. Epub 2019 Jul 17. PMID 31315940